CLINICAL TRIAL: NCT01147770
Title: The Effect of Progesterone Supplementation During Early Gestations in Patients Treated With Rec FSH/GnRH Antagonist:a Randomized Controlled Trial
Brief Title: Prolongation of Progesterone Supplementation in Antagonist Cycles and Pregnancy Outcomes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Kyrou Dimitra, Resident, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRG-45
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Infertility
Keywords: progesterone; antagonist; rec FSH; IVF; pregnancy
MeSH Terms: conditions — Infertility | interventions — Progesterone; Utrogestan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stop progesterone (Experimental)
  Interventions: Drug: progesterone

INTERVENTIONS:
Drug: progesterone — duration
  Other Names: utrogestan

SUMMARY:
The objective of this study is to evaluate the effect of the prolongation of luteal support on the ongoing pregnancy rate (beyond 12 weeks of gestation )in recFSH/GnRH antagonist cycles.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or less than 39
* Body mass index between 18-29 kg/m2
* Presence of both ovaries
* Basal hormonal values on day 2 of the cycle
* Embryotransfer day3 or day5
* 1 to 3 cycles

Exclusion Criteria:

* Endometriosis stage 3
* Polycystic ovarian syndrome
* Frozen or testicular sperm

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2008-09; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy rate | up to 2 years